CLINICAL TRIAL: NCT00939120
Title: A Randomized, Double-blind, Placebo-controlled, Study of Safety and Efficacy of Dutasteride in Combination With Tolterodine ER or Placebo in Men With Lower Urinary Tract Symptoms (LUTS) Including Urgency and Frequency
Brief Title: Dutasteride With Tolterodine ER or Placebo to Treat Lower Urinary Tract Symptoms (LUTS)
Acronym: LUTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Siami, Paul F., M.D. (Other)
Collaborators: GlaxoSmithKline (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Paul F. Siami, MD, Medical Director, Deaconess Clinic Research Institute, Siami, Paul F., M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110983
Record Dates: First submitted 2009-06-12; First posted 2009-07-14 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign prostatic hyperplasia (BPH); dutasteride; tolterodine ER
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolterodine ER 4mg (Experimental): 1:1 randomization to either Dutasteride 0.5mg orally once daily plus Tolterodine ER 4mg orally once daily or Dutasteride 0.5mg orally once daily plus placebo once daily
  Interventions: Drug: Tolterodine ER 4mg; Drug: Pre-randomization Dutasteride
- placebo (Placebo Comparator): 1:1 randomization to either Dutasteride 0.5mg orally once daily plus Tolterodine ER 4mg orally once daily or Dutasteride 0.5mg orally once daily plus placebo once daily
  Interventions: Drug: Placebo; Drug: Pre-randomization Dutasteride

INTERVENTIONS:
Drug: Tolterodine ER 4mg — 1:1 randomization to either Dutasteride 0.5mg orally once daily plus Tolterodine ER 4 mg orally once daily or Dutasteride 0.5mg orally once daily plus placebo once daily
  Other Names: Detrol LA
  Arms: Tolterodine ER 4mg
Drug: Placebo — 1:1 randomization to either Dutasteride 0.5mg orally once daily plus Tolterodine ER 4mg orally once daily or Dutasteride 0.5mg orally once daily plus placebo once daily
  Arms: placebo
Drug: Pre-randomization Dutasteride — All participants were on Dutasteride 0.5mg orally once daily prior to randomization.

SUMMARY:
This is an investigator-initiated study of safety, efficacy and tolerability of dutasteride given for 18 months, including a 1-year double-blind randomized co-administration with either tolterodine ER or placebo in men suffering from lower urinary tract symptoms (LUTS) including urgency and frequency, with or without urgency urinary incontinence (i.e., overactive bladder (OAB) symptoms).

DETAILED DESCRIPTION:
Men who are treated with an alpha blocker (AB) or 5-alpha reductase inhibitor (5-ARI) for benign prostatic enlargement (BPE) and lower urinary tract symptoms (LUTS) often have symptoms including urinary frequency and urgency. ABs and 5-ARIs may improve the obstructive voiding symptoms but not necessarily the storage symptoms.

This study will evaluate the safety and efficacy of dutasteride 0.5 mg once daily for 6 months in an open label fashion. Those patients who continue to report storage urinary symptoms, will be randomized to receive dutasteride 0.5 mg once daily for an additional one year together with double-blind tolterodine ER 4 mg or matched tolterodine ER placebo once daily.

ELIGIBILITY:
Inclusion Criteria:

This subject population will consist of males ≥ 50 years of age who have lower urinary tract symptoms (LUTS) due to benign prostatic enlargement (BPE) for a minimum of 3 months

Inclusion criteria at screening:

1. Subjects who understand and speak English and are able to comply with the protocol, complete the diaries, and other study tools
2. Subject has provided written informed consent and HIPAA authorization
3. Ambulatory male subjects ≥ 50 years of age
4. Able to use the toilet without difficulty
5. History of LUTS due to BPE, as diagnosed by history as well as digital rectal exam (DRE), for ≥ 3 months suitable for medical therapy with 5-ARI in combination with antimuscarinic drugs
6. Prostate volume (PV) ≥ 30 cc as measured by transrectal ultrasound (TRUS)
7. International prostate symptoms score (IPSS) ≥12
8. Post Void Residual Volume < 150 mL at baseline
9. Uroflowmetry-Qmax > 5 mL/sec and ≤ 15 mL/sec
10. Prostate specific antigen (PSA) ≥ 1.5 ng/ml and in normal age-adjusted range. For those subjects with an elevated age-adjusted PSA, it is the responsibility of the investigator to take standard of care measures to assure reasonable absence of prostate cancer
11. Have an average of ≥ 8 micturitions per 24 hrs
12. Have an average of 2 episodes of urgency per 24 hrs (defined as those with the Urinary Sensation Scale rating of 3 or more)

Exclusion Criteria:

1. Concurrent use of 5-ARI therapy within the past 3 months
2. Concurrent use of alpha blockers within the past 2 weeks
3. Concurrent use of antimuscarinics within the past 4 weeks
4. Concurrent use of Phosphodiesterase type 5 (PDE-5) inhibitors on a daily basis
5. Evidence of chronic inflammation such as interstitial cystitis and bladder stones.
6. Evidence of untreated urethral stricture disease
7. Uncontrolled narrow angle glaucoma
8. Increased post-void residual volume (PVR) defined as PVR > 150 mL
9. Uroflowmetry-Qmax ≤ 5 mL/sec
10. Acute urinary tract infection (UTI). These subjects may be treated and re-screened
11. Acute urinary retention (AUR) requiring catheter within the last 3 months
12. Previous or planned transurethral resection of the prostate (TURP)
13. Minimally invasive surgery (MIS) such as transurethral microwave treatment (TUMT), transurethral needle ablation (TUNA), laser, or other minimally invasive procedures within 12 months. Those patients who in the opinion of the investigator did not respond adequately to MIS and fulfill the inclusion criteria are eligible to participate
14. A known diagnosis of prostate cancer.
15. A known diagnosis of bladder cancer within 5 years of screening. Those patients with history of non-muscle invasive bladder cancer who have not had a recurrence in the past 5 years are eligible to screen for this study and must maintain continued adequate bladder cancer screening at the discretion of the Investigator
16. Renal or hepatic impairment defined as 2.5 x upper limit of normal. Some isolated abnormalities would be left at the discretion of the investigator with always keeping in mind to not pose a hazard to the patient.
17. PSA > 10 ng/mL (if the PSA is greater than 4 ng/mL and less than or equal to 10 ng/mL, subjects may be included at the discretion of the Investigator if the PSA has been stable and the patient has had a prostate biopsy showing no evidence of prostate cancer)
18. Known or suspected hypersensitivity to dutasteride or tolterodine ER .
19. Participation in a clinical trial involving an investigational drug, within 30 days prior to enrollment.
20. History of diagnosed gastrointestinal obstruction disease.
21. Myocardial infarction within the past 8 weeks.
22. Known or suspected drug and/or alcohol abuse.
23. Any clinical condition, which, in the opinion of the Investigator, would not allow safe completion of the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Siami, MD, Principal Investigator — Deaconess Clinic Research Institute
Locations (1):
- Deaconess Clinic Gateway Health Center, Newburgh, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolterodine ER 4mg + Dutasteride 0.5mg: Patients randomized to experimental group received Dutasteride 0.5mg orally once daily plus Tolterodine ER 4mg orally once daily.
- Placebo + Dutasteride 0.5mg: Patients randomized to control group received Dutasteride 0.5mg orally once daily plus placebo orally once daily.
Period: Overall Study
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Started | 23 | 23
Completed | 15 | 18
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Population: Number of patients randomized into control or experimental groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of patient at enrollment
  years | 68.6 (9.5) | 67.7 (7.4) | 68.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of participant.
  Participants
    Female | 0 | 0 | 0
    Male | 23 | 23 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of the participant.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 23 | 22 | 45
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Region in which participant was enrolled.
  participants
    United States | 23 | 23 | 46
Prostate volume [Mean (Standard Deviation); unit: mL] — Prostate volume measured by transrectal ultrasound, age-adjusted for this study.
  mL | 43.9 (15.8) | 43.1 (16.0) | 43.5 (15.7)
Prostate specific antigen [Mean (Standard Deviation); unit: ng/mL] — Prostate specific antigen measured via blood test.
  ng/mL | 4.0 (2.1) | 5.3 (8.8) | 4.6 (6.4)
Voided volume [Mean (Standard Deviation); unit: mL] — Voided urinary volume via uroflowmetry.
  mL | 202.5 (96.5) | 273.7 (189.9) | 238.1 (153.2)
Maximum flow rate [Mean (Standard Deviation); unit: mL/sec] — Maximum urine flow rate (Qmax) measured via uroflowmetry.
  mL/sec | 11.1 (3.5) | 12.4 (4.8) | 11.7 (4.2)
Post-void residual volume [Mean (Standard Deviation); unit: mL] — Post-voiding residual volume (PVR) measured in each participant via ultrasound.
  mL | 93.0 (69.2) | 81.6 (60.7) | 87.3 (64.6)
Overactive bladder questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Overactive Bladder Questionnaire score is based on the answers to 33 questions concerning bladder symptoms. Each question is assigned points from 1 to 6 indicating increasing severity of the particular symptom. The total score can therefore range from 33 to 198 (asymptomatic to very symptomatic).
  units on a scale | 86.4 (22.3) | 86.1 (29.9) | 86.3 (26.1)
Patient's perception of bladder condition [Mean (Standard Deviation); unit: units on a scale] — Patient-reported scores on a scale of 1-6 indicating how their bladder condition affects them. Scores are as follows: 1 = Does not cause me any problems at all; 2 = Causes me some very minor problems; 3 = Causes me some minor problems; 4 = Causes me (some) moderate problems; 5 = Causes me severe problems; 6 = Causes me many severe problems.
  units on a scale | 3.7 (0.9) | 3.7 (1.0) | 3.7 (0.9)
International prostate symptoms score, total [Mean (Standard Deviation); unit: units on a scale] — The IPSS is based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  units on a scale | 18.0 (6.2) | 17.7 (4.5) | 17.9 (5.4)
International prostate symptoms score, voiding subscore [Mean (Standard Deviation); unit: units on a scale] — The IPSS is based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  Voiding sub-component is 4/7 questions, thus ranging from 0-20.
  units on a scale | 9.1 (4.3) | 9.0 (3.8) | 9.1 (4.0)
International prostate symptoms score, storage subscore [Mean (Standard Deviation); unit: units on a scale] — The IPSS is based on the answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  Storage sub-component is 3/7 questions, thus ranging from 0-15.
  units on a scale | 8.9 (2.7) | 8.7 (2.2) | 8.8 (2.4)
Urinary urgency [Mean (Standard Deviation); unit: urgency episodes] — Patient reported number of urgency episodes during a 24-hour period.
  urgency episodes | 6.7 (3.5) | 8.6 (3.5) | 7.7 (3.6)
Urinary frequency [Mean (Standard Deviation); unit: frequency episodes] — Participant reported urinary frequency episodes during a 24-hour period.
  frequency episodes | 11.3 (2.2) | 11.4 (2.2) | 11.3 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Post-void Residual (PVR) Volume
Description: To evaluate the safety of dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with symptoms of LUTS: post-voiding residual volume measured via ultrasound.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: mL
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
mL | 101.7 (22.4) | 75.8 (9.6)

2. Secondary Outcome: Overactive Bladder Questionnaire (OABq)
Description: To evaluate the efficacy in men taking dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with LUTS including OAB symptoms: overactive bladder questionnaire (OABq) - 33 questions scored via 1-6 (higher scores indicate more severe symptoms), thus values ranged from 33-198.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
units on a scale | 80.2 (5.8) | 67.7 (5.3)

3. Primary Outcome: Maximum Urine Flow Rate (Qmax).
Description: To evaluate the safety of dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with symptoms of LUTS: maximum urine flow rate (Qmax) measured via uroflowmetry.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: mL/sec
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
mL/sec | 11.7 (0.7) | 12.9 (1.7)

4. Primary Outcome: Urine Voided Volume (Voiding)
Description: To evaluate the safety of dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with symptoms of LUTS: urine voided volume (voiding) measured by uroflowmetry.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: mL
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
mL | 219.9 (20.6) | 232.9 (32.3)

5. Primary Outcome: Acute Urinary Retention (AUR)
Description: To evaluate the safety of dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with symptoms of LUTS: acute urinary attention (AUR) - inability to urinate requiring catheterization.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Number; unit: participants
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
participants | 0 | 0

6. Secondary Outcome: Patient Perception of Bladder Condition (PPBC)
Description: To evaluate the efficacy in men taking dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with LUTS including OAB symptoms: participant reported patient perception of bladder condition (PPBC), one question scored from 1-6, higher scores indicating more severe symptoms.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
units on a scale | 3.6 (0.3) | 3.0 (0.2)

7. Secondary Outcome: International Prostate Symptoms Score (IPSS), Total
Description: To evaluate the efficacy in men taking dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with LUTS including OAB symptoms: total international prostate symptoms score (IPSS) - 7 questions scored from 0-5 (higher score indicating more severe symptoms), thus total scores ranged from 0-35.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
units on a scale | 15.4 (1.4) | 14.5 (1.3)

8. Secondary Outcome: International Prostate Symptoms Score, Voiding Subscore
Description: To evaluate the efficacy in men taking dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with LUTS including OAB symptoms: voiding subscore of international prostate symptoms score (IPSS) - 4 questions scored from 0-5 (higher score indicating more severe symptoms), thus total scores ranged from 0-20.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
units on a scale | 7.5 (1.0) | 7.0 (0.9)

9. Secondary Outcome: International Prostate Symptoms Score (IPSS), Storage Subscore
Description: To evaluate the efficacy in men taking dutasteride 0.5 mg in combination with either tolterodine ER 4mg or placebo for the treatment of men with LUTS including OAB symptoms: storage subscore international prostate symptoms score (IPSS) - 3 questions scored from 0-5 (higher score indicating more severe symptoms), thus total scores ranged from 0-15.
Time Frame: 12 months
Population: Last data point carried forward for participants who were randomized and dropped prior to study end.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Number analyzed (Participants) | 23 | 23
units on a scale | 7.9 (0.7) | 7.5 (0.6)

ADVERSE EVENTS:
Time Frame: 19 months.
Description: Reported all adverse events broken up based on categorization as adverse event, serious adverse event, and possibly drug-related adverse event.
Arm/Group | Tolterodine ER 4mg + Dutasteride 0.5mg | Placebo + Dutasteride 0.5mg
Serious Adverse Events (participants affected / at risk) | 4/23 | 5/23
Other Adverse Events (participants affected / at risk) | 21/23 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolterodine ER 4mg + Dutasteride 0.5mg (N=23) | Placebo + Dutasteride 0.5mg (N=23)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0) — Moderate, intermittent
Nasal airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Bilateral, moderate intensity.
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Mild intensity
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0) — Severe
Gallstones (Hepatobiliary disorders) | 0 (0) | 1 (1) — Severe, requiring cholecystectomy
Mass on kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Severe, continuous.
Cervical stenosis (Nervous system disorders) | 0 (0) | 1 (1) — Severe
Oral thrush (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild
Schatzki ring (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild, continuous, shallow
Presbyesophagus, dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Moderate to severe
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Severe, continuous
Hiatal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild, continuous
Suicidal self-inflicted gunshot wound, lethal (Psychiatric disorders) | 0 (0) | 1 (1)
Gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Moderate intermittent exacerbation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolterodine ER 4mg + Dutasteride 0.5mg (N=23) | Placebo + Dutasteride 0.5mg (N=23)
Epistaxis (Blood and lymphatic system disorders) | 2 | 0
Difficulty urinating (Renal and urinary disorders) | 3 | 2
Urinary urgency / incontinence (Renal and urinary disorders) | 5 | 2
URI / sinusitis / rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Otitis media (Ear and labyrinth disorders) | 2 | 1
Bronchitis / pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 4
Actinic keratosis, basal cell carcinoma (Skin and subcutaneous tissue disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Increase in prostate specific antigen (Reproductive system and breast disorders) | 2 | 0
Prostate nodule (Reproductive system and breast disorders) | 2 | 0
Cataracts (Eye disorders) | 0 | 3 — Incidence and surgery of cataracts
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Fatigue (General disorders) | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 2
Groin pain (Reproductive system and breast disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Angina (Cardiac disorders) | 0 | 2
Diabetes (Endocrine disorders) | 1 | 2
Kidney stones (Renal and urinary disorders) | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Gynecomastia (Reproductive system and breast disorders) | 1 | 3
Breast tenderness (Reproductive system and breast disorders) | 4 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No